CLINICAL TRIAL: NCT02057705
Title: Prospective, Longitudinal Study of the Natural History and Functional Status of Patients With Myotubular Myopathy (MTM)
Acronym: MTM
Status: Completed | Type: Observational
Sponsor: Valerion Therapeutics, LLC (Industry)
Collaborators: Institut de Myologie, France (Other); Genethon (Other)
Responsible Party: Sponsor
Other Study IDs: VAL-101-13
Record Dates: First submitted 2014-02-04; First posted 2014-02-07 (Estimated); Last update posted 2018-06-07 (Actual); Status verified 2018-06

CONDITIONS: Myotubular Myopathy
Keywords: MTM; myotubular myopathy; X-linked centronuclear myopathy; inherited myopathies; neuromuscular diseases; hypotonia; genetic mutation
MeSH Terms: conditions — Myopathies, Structural, Congenital; Neuromuscular Diseases; Muscle Hypotonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * 5 ml sample of whole blood will be collected during the study to assess the immunity against various AAV serotypes
  * 5 ml blood sample may be obtained for peripheral blood mononuclear cells (PBMC) to quantify X-linked myotubular myopathy gene 1 (MTM1) production
  * 24-hour urine collection will be performed every 6 months in order to measure urinary creatinine excretion
  * Slides and tissue from a previously performed muscle biopsy will be obtained for a central review and quantification of histo- and immunohistopathological features of MTM
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a prospective, non-interventional, longitudinal study of the natural history and function of approximately 60 patients with MTM from the United States, Canada and Europe. The duration of the study, including the enrollment period, will be 36 months. Data from the study will be used to characterize the disease course of MTM and determine which outcome measures will be the best to assess the efficacy of potential therapies.

DETAILED DESCRIPTION:
This is a prospective, non-interventional, longitudinal study of the natural history and function of patients with MTM. The study duration is 36 months. The enrollment period will be 12 months and each patient will be assessed over 24 months. Data will be analyzed at baseline and annually thereafter and reports will be prepared based on these analyses. A final report will summarize findings after all patients have completed 24 months of follow-up. Assessments performed in this study will be based on the age and ambulatory status of the patient. The assessments will also be adjusted to account for the variability in both phenotypes and age of the patients who may participate in this study. Patients will be evaluated at Baseline, Month 6, Month 12 and Month 24. It is anticipated that approximately 60 patients from the United States, Canada and Europe will be included in this study.

ELIGIBILITY:
Inclusion criteria:

* Patients of any age (newborns included) may participate.
* Patients over 18 years of age and parent(s)/legal guardian(s) of patients <18 years of age must provide written informed consent prior to participating in the study and informed assent will be obtained from minors at least 7 years of age when required by regulation.
* MTM resulting from a mutation in the MTM1 gene.
* Male or symptomatic female. A symptomatic female will be defined by the motor function assessment by Motor Function Measure (MFM) or North Star Ambulatory Assessment (NSAA) below 80% of the total score.
* Willing and able to comply with all protocol requirements and procedures.

Exclusion criteria:

* Other disease which may significantly interfere with the assessment of MTM and is clearly not related to the disease.
* Currently enrolled in a treatment study; or treatment with an experimental therapy other than pyridostigmine.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Investigative Research Centers
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2014-02; Primary Completion 2017-06-26 (Actual); Study Completion 2017-06-26 (Actual)

PRIMARY OUTCOMES:
Time to characterize the disease course in MTM patients | Up to 24 Months
  Study-specific functional assessments and patient questionnaires will be used and will be based on the age and ambulatory status of the participant

SECONDARY OUTCOMES:
Change in disease severity and disease progression | Baseline, Month 3 (EU only), Month 6, Month 12 and Month 24
  Study-specific functional assessments and patient questionnaires will be used and will be based on the age and ambulatory status of the participant

OTHER OUTCOMES:
Number of participants with an immune response against adeno-associated virus (AAV) | Baseline Visit
  A 5 ml sample of whole blood will be collected during the study to assess the immunity against various AAV serotypes.

CONTACTS AND LOCATIONS:
Overall Officials: Hal Landy, MD, Study Director — Valerion Therapeutics, LLC
Locations (13):
- Boston Children's Hospital, 300 Longwood Avenue, Boston, Massachusetts, United States
- Centre Hospitalier Regional de la Citadelle, Liège, Belgium
- Hospital for Sick Children, 555 University Avenue, Toronto, Ontario, Canada
- France (7):
  - Hôpital Femme Mère Enfant, CHU Lyon Escale, Bron
  - Roger Salengro Hospital, CHU, Lille, Lille
  - Croix Rousse Hospital, Lyon
  - Hôpital Armand Trousseau, Paris
  - Institut I-Motion, Hôpital A. Trousseau, Paris
  - Institut de Myologie, GH Pitié Salpêtrière, Bâtiment Babinski, Paris
  - Hôpital Sainte Musse, Toulon
- University Hospital of Essen, Essen, Germany
- Bambino Gesù Children's Hospital, Rome, Italy
- Hôpital Puertas de Mar, Cadiz, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Herman GE, Finegold M, Zhao W, de Gouyon B, Metzenberg A. Medical complications in long-term survivors with X-linked myotubular myopathy. J Pediatr. 1999 Feb;134(2):206-14. doi: 10.1016/s0022-3476(99)70417-8. PMID 9931531
- [Background] Jungbluth H, Sewry CA, Buj-Bello A, Kristiansen M, Orstavik KH, Kelsey A, Manzur AY, Mercuri E, Wallgren-Pettersson C, Muntoni F. Early and severe presentation of X-linked myotubular myopathy in a girl with skewed X-inactivation. Neuromuscul Disord. 2003 Jan;13(1):55-9. doi: 10.1016/s0960-8966(02)00194-3. PMID 12467733
- [Background] McEntagart M, Parsons G, Buj-Bello A, Biancalana V, Fenton I, Little M, Krawczak M, Thomas N, Herman G, Clarke A, Wallgren-Pettersson C. Genotype-phenotype correlations in X-linked myotubular myopathy. Neuromuscul Disord. 2002 Dec;12(10):939-46. doi: 10.1016/s0960-8966(02)00153-0. PMID 12467749
- [Background] Jungbluth H, Wallgren-Pettersson C, Laporte J. Centronuclear (myotubular) myopathy. Orphanet J Rare Dis. 2008 Sep 25;3:26. doi: 10.1186/1750-1172-3-26. PMID 18817572
- [Derived] Annoussamy M, Lilien C, Gidaro T, Gargaun E, Che V, Schara U, Gangfuss A, D'Amico A, Dowling JJ, Darras BT, Daron A, Hernandez A, de Lattre C, Arnal JM, Mayer M, Cuisset JM, Vuillerot C, Fontaine S, Bellance R, Biancalana V, Buj-Bello A, Hogrel JY, Landy H, Servais L. X-linked myotubular myopathy: A prospective international natural history study. Neurology. 2019 Apr 16;92(16):e1852-e1867. doi: 10.1212/WNL.0000000000007319. Epub 2019 Mar 22. PMID 30902907
- See also: National Institute of Health — http://ghr.nlm.nih.gov/condition/x-linked-myotubular-myopathy
- See also: Muscular Dystrophy Association — https://www.mda.org/disease/inherited-and-endocrine-myopathies